CLINICAL TRIAL: NCT05797363
Title: The Effect of Continuous Midwife Support During Pregnancy, Childbirth and Postpartum Processes Starting From Preconceptional Period on Various Parameters Related to Pregnancy, Delivery and Postpartum Period: A Randomized Controlled Study"
Brief Title: The Effect of Continuous Midwife Support on Various Parameters Related to Pregnancy, Childbirth and Postpartum Period
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AmasyaU-1
Record Dates: First submitted 2021-09-20; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Pregnant Women; Childbirth; Women's Health

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Experimental): Continuous midwifery support will be applied to the intervention group. The women included in the experimental group will be counseled on many issues such as nutrition, vaccinations, family planning, pregnancy follow-ups, normal birth and cesarean section surgery, coping with labor pain, puerperium process, baby care, starting from the pre-pregnancy period, during pregnancy, childbirth and postpartum periods.
  Interventions: Other: Continuous midwife support
- Control Group (No Intervention): No action will be taken against this group.

INTERVENTIONS:
Other: Continuous midwife support — The individuals included in the experimental group will be provided with consultancy services on many issues from the pre-pregnancy period to the postpartum period.
  Arms: Experiment

SUMMARY:
There is a need for studies with a high level of evidence regarding the effect of supportive care given during the preconceptional period, pregnancy, childbirth and postpartum processes. With this planned study, it is aimed to evaluate the effect of continuous midwife support during pregnancy, birth and postpartum periods, starting from the preconceptional period, on various parameters related to pregnancy, birth and postpartum period. The research is planned as a randomized controlled experimental study. It consists of two groups, the study group and the control group. 75 women out of 150 women will form the control group and 75 women will form the study group. The women in the working group will be given individual training in line with their needs. Data will be collected by using the checklist and many scales used by the control and study groups in preconceptional counseling recommended by ACOG (American College of Obstetricians and Gynecologists).

DETAILED DESCRIPTION:
INTRODUCTION Globally, midwives are the primary caregivers of women during pregnancy, childbirth, and postpartum. It is recommended to use a midwife-led care model to provide support and assistance to women during pregnancy, childbirth, and the postpartum period. In midwife-led care, midwifery provides quality health care services to women and newborns during pregnancy, delivery, and the postpartum period. Therefore, the evidence-based literature from developed and developing countries emphasizes that maternal and neonatal mortality can be reduced with midwife-led care. Studies suggest that the constant presence of midwives during pregnancy, childbirth, and postpartum period encourages women. Continuity of care increases women's trust in midwives.

In the literature, no study has been found in which the effect of midwifery care initiated in the preconceptional period on pregnancy, birth or postpartum processes has been investigated. For this reason, it is thought that the research will provide meaningful data to the literature.

METHOD

The research is planned as a randomized controlled experimental study. Randomization is planned to be done by the second researcher in a computer environment using the www.randomizer.org internet address. Women numbered 1-150 will be assigned to the study and control groups. The assignment of women to the groups, analysis, and reporting stages will be done by the second researcher, and data collection, training, and follow-up will be done by the first and third researchers. Thus, data collection, training, and follow-up for the second researcher, and the assignment of women to the group for the first and third researcher, analysis, and reporting will be blinded. It consists of two groups, the study group, and the control group. 150 women who applied to Family Health Centers to get a health report for marriage and agreed to participate in the study will be identified. 75 women out of 150 women will form the control group and 75 women will form the study group. The control list used in preconception counseling recommended by ACOG (American College of Obstetricians and Gynecologists) and the scales will be used by both the control and study groups. The pregnancy, delivery, and postpartum period processes of 150 women will be followed starting from the preconception period. 75 women will be given training in line with their individual needs. 75 women will not be given any training. The data will be analyzed using the SPSS package program. Appropriate statistical analysis tests will be used in the analysis of the data by looking at the normality distribution.

Intervention group

1. Meeting- Preconception ACOG Preconception Counseling Checklist and personal information form
2. Meeting- Preconception Education
3. Meeting- Preconception Education and the Childbirth Fear - Prior to Pregnancy Scale and family planning scale
4. Meeting (First Trimester in Pregnancy) Education in pregnancy
5. Meeting (First Trimester in pregnancy) Education in pregnancy and Health Practices Questionnaire In Pregnancy
6. Meeting (First Trimester in pregnancy) Education and the scale of Self-perception of Pregnants, Pregnancy Experience Scale (PES)
7. Meeting (Second Trimester in pregnancy) Education and Perception of Pregnancy Risk Scale
8. Meeting (Second Trimester in pregnancy) Education and Pregnancy-related Anxiety Scale
9. Meeting (Third Trimester in pregnancy) Education and Pregnancy Experience Scale, Prenatal Care Satisfaction Scale
10. Meeting (Third Trimester in pregnancy) "Education and Prenatal Breastfeeding Self-Efficacy Scale, Health Practices Questionnaire in Pregnancy-II"
11. Meeting (Third Trimester in pregnancy) Education and Scale of Childbirth of Self Efficacy, Antenatal Perceived Stress Scale, The Oxford Worries About Labour Scale
12. Meeting ( Labour) "Education- supportive and Scale Of Woman's Perception Of Supportive Care Given To Woman In Labor, Partograph, the Childbirth Comfort Questionnaire"
13. Meeting (Postpartum - first day) Postpartum follow-up breastfeeding support
14. Meeting (Postpartum - 1-7 days) Postpartum follow-up, education
15. Meeting (Postpartum - 7-21 days) Postpartum follow-up, education
16. Meeting (Postpartum - 30-42 days) "Education and Maternal Postpartum Quality of Life Questionnaire, the Mothers' Postnatal Sense of Security Scale and Postpartum Sleep Quality Scale

Control Group

1. Meeting- Preconception ACOG Preconception Counseling Checklist and personal information form
2. Meeting- Preconception
3. Meeting- Preconception the Childbirth Fear - Prior to Pregnancy Scale and family planning scale
4. Meeting (First Trimester in Pregnancy)
5. Meeting (First Trimester in pregnancy) Health Practices Questionnaire In Pregnancy
6. Meeting (First Trimester in pregnancy) the scale of Self-perception of Pregnants, Pregnancy Experience Scale (PES)
7. Meeting (Second Trimester in pregnancy) Perception of Pregnancy Risk Scale
8. Meeting (Second Trimester in pregnancy) Pregnancy-related Anxiety Scale
9. Meeting (Third Trimester in pregnancy) Pregnancy Experience Scale, Prenatal Care Satisfaction Scale
10. Meeting (Third Trimester in pregnancy) " Prenatal Breastfeeding Self-Efficacy Scale, Health Practices Questionnaire in Pregnancy-II"
11. Meeting (Third Trimester in pregnancy) Scale of Childbirth of Self Efficacy, Antenatal Perceived Stress Scale, The Oxford Worries About Labour Scale
12. Meeting ( Labour) "Scale Of Woman's Perception Of Supportive Care Given To Woman In Labor, Partograph, the Childbirth Comfort Questionnaire"
13. Meeting (Postpartum - first day)
14. Meeting (Postpartum - 1-7 days)
15. Meeting (Postpartum - 7-21 days)
16. Meeting (Postpartum - 30-42 days) "Maternal Postpartum Quality of Life Questionnaire, the Mothers' Postnatal Sense of Security Scale and Postpartum Sleep Quality Scale "

ELIGIBILITY:
Inclusion Criteria:

* She's newly married.
* Women without children.

Exclusion Criteria:

* women's desire to stop working

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-04-15 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Perception of Pregnancy Risk Scale (PPRS) | average of 1 year
  PPRS: An increase in the score obtained from the scale is interpreted as an increase in the risk perception of the pregnant woman and her baby.
Pregnancy-related Anxiety Scale (PrAS) | average of 1 year
  PrAS: The cut-off score calculated for the scale is 75.5. A total score of 75.5 and above indicates an increased anxiety level due to pregnancy.
CHILDBIRTH FEAR - PRIOR TO PREGNANCY SCALE (CFPPS) | average of 1 year
  CFPPS: While the minimum score on the scale is 10, the maximum score is 60. A high item total score indicates a high level of fear.
Antenatal Perceived Stress Scale (APSS) | average of 1 year
  APSS: The perceived stress score during pregnancy is obtained by summing the item scores in the scale and then dividing by the number of items. While the lowest score that can be obtained from the scale is 1, the highest score is 5. The high total score obtained from the scale indicates the highest perceived stress level in pregnant women.
Prenatal breastfeeding self efficacy scale (PBSeS) | average of 1 year
  PBSeS: Each item of the scale is graded as a 5-point Likert type. The lowest score that can be obtained from the total of the scale is 20, and the highest score is 100. The higher the score, the higher the perception of breastfeeding self-efficacy.
Family Planning Attitude Scale (FPAS) | average of 1 year
  FPAS: The scale is a five-point Likert-type scale consisting of 34 items. The lowest 34 and the highest 170 points can be obtained from the scale, and an increase in the total score means a more positive family planning attitude.
Prenatal Care Satisfaction Scale (PCSS) | average of 1 year
  PCSS: There is no cut-off point in the evaluation of the scale. The higher the score obtained from the scale, the higher the satisfaction, and the lower it is, the lower the satisfaction.
Oxford Birth Anxiety Scale (OBAS) | average of 2 year
  OBAS: The scale is evaluated over the total score (min=10, max=40). As the score increases, it is interpreted that the anxiety level of women increases.
Pregnancy Experience Scale (PES) | average of 2 year
  PES: A total of six sub-dimension scores (positive emotions frequency score, negative emotions frequency score, positive emotions intensity score, negative emotions intensity score, frequency ratio and intensity ratio) are obtained in GDS.
Self-perception of Pregnants Scale (SPS) | average of 2 year
  SPS: When evaluating the scores of the Pregnancy Body Perception sub-dimension, high scores indicate negative pregnancy body perception, and low scores indicate positive pregnancy body perception. The highest score that can be obtained in the Pregnancy Body Perception sub-dimension is 20, and the lowest score is 5.
HEALTH PRACTICES QUESTIONNAIRE IN PREGNANCY | average of 2 year
  The highest score that can be obtained from the scale is 165, and the lowest score is 33. High scores indicate good health practices.
Childbirth Comfort Questionnaire (CCQ) | average of 3 year
  CCQ: The minimum score that can be obtained from the scale is 14, the highest score is 70. As the score increases, it is said to be high-level comfort, and as the score decreases, low-level comfort is mentioned.
MOTHERS' POSTNATAL SENSE OF SECURITY SCALE (MPSSS) | average of 3 year
  MPSSS: Scores from the scale range from 18 to 72, and high scores indicate good feelings of security.
Postpartum Quality of Life Questionnaire (PQLQ) | average of 3 year
  PQLQ: The higher the score obtained from the scale, the higher the person's postpartum quality of life, and lower scores the lower the postpartum quality of life.
SCALE OF WOMAN'S PERCEPTION OF SUPPORTIVE CARE GIVEN TO WOMAN IN LABOR | average of 3 year
  At least 33 from the scale; maximum 132 points are taken. There is no cut-off point in the scale. The higher the score from the scale, the better the supportive nursing care received.
Childbirth Self-Efficacy Scale (CSES) | average of 3 year
  CSES: The lowest total score that can be obtained from the scale is 32, and the highest total score is 320. High scores from the scale show that pregnant women have high self-efficacy levels in labor.
Postpartum Sleep Quality Scale (PSQS) | average of 3 year
  PSQS: The lowest 0 and the highest 56 points can be obtained from the scale and there is no cut-off point. An increase in the score indicates a decrease in sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: duygu murat, öztürk, Study Director — duygu.murat@hotmail.com

IPD SHARING:
Plan to Share IPD: Yes
The data obtained is planned to be published as a scientific article.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: up to 6 years